CLINICAL TRIAL: NCT06122805
Title: Effectiveness of Dual Light Therapy Electric Toothbrush vs.Manual Toothbrush on Periodontal Health of Orthodontic Patients Undergoing Oral Surgery
Brief Title: Effectiveness of Dual Light Electric Toothbrush vs. Manual Toothbrush in Orthodontic Patients Undergoing Oral Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Los Angeles (Other)
Responsible Party: Principal Investigator, Stephen Yen, Associate Professor, Children's Hospital Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CHLA-23-00184
Record Dates: First submitted 2023-11-03; First posted 2023-11-08 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Toothbrushing; Gingivitis; Cleft Lip and Palate
MeSH Terms: conditions — Gingivitis; Cleft Lip

STUDY DESIGN:
Intervention Model Description: Randomized
Who Masked: Investigator
Masking Description: randomized assignment of study ID number
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (9):
- Orthognathic Surgery Manual Toothbrush (Experimental): 1. Patient of record of the Craniofacial and Special Care Orthodontic Clinic at Children's Hospital Los Angeles
  2. Between the ages of 6 and 20 years
  3. Physical status of ASA I or II
  4. Diagnosis of craniofacial and/or isolated, complete or incomplete, bilateral or unilateral cleft lip and palate
  5. Intervention: Manual toothbrush.
  Interventions: Device: Toothbrush
- Orthognathic Surgery Sonic toothbrush (Experimental): 1. Patient of record of the Craniofacial and Special Care Orthodontic Clinic at Children's Hospital Los Angeles
  2. Between the ages of 6 and 20 years
  3. Physical status of ASA I or II
  4. Diagnosis of craniofacial and/or isolated, complete or incomplete, bilateral or unilateral cleft lip and palate
  5. Intervention:Sonic toothbrush without activation of the dual light feature.
  Interventions: Device: Toothbrush
- Orthognathic Surgery Sonic and dual light toothbrush (Experimental): 1. Patient of record of the Craniofacial and Special Care Orthodontic Clinic at Children's Hospital Los Angeles
  2. Between the ages of 6 and 20 years
  3. Physical status of ASA I or II
  4. Diagnosis of craniofacial and/or isolated, complete or incomplete, bilateral or unilateral cleft lip and palate
  5. Intervention:Sonic toothbrush with activation of the dual light feature
  Interventions: Device: Toothbrush
- Bone Graft Manual Toothbrush (Experimental): 1. Patient of record of the Craniofacial and Special Care Orthodontic Clinic at Children's Hospital Los Angeles
  2. Between the ages of 6 and 20 years
  3. Physical status of ASA I or II
  4. Diagnosis of craniofacial and/or isolated, complete or incomplete, bilateral or unilateral cleft lip and palate
  5. Intervention:Manual toothbrush.
  Interventions: Device: Toothbrush
- Bone Graft Sonic Toothbrush (Experimental): 1. Patient of record of the Craniofacial and Special Care Orthodontic Clinic at Children's Hospital Los Angeles
  2. Between the ages of 6 and 20 years
  3. Physical status of ASA I or II
  4. Diagnosis of craniofacial and/or isolated, complete or incomplete, bilateral or unilateral cleft lip and palate
  5. Intervention:Sonic toothbrush without activation of the dual light feature.
  Interventions: Device: Toothbrush
- Bone Graft Sonic and Dual-light Toothbrush (Experimental): 1. Patient of record of the Craniofacial and Special Care Orthodontic Clinic at Children's Hospital Los Angeles
  2. Between the ages of 6 and 20 years
  3. Physical status of ASA I or II
  4. Diagnosis of craniofacial and/or isolated, complete or incomplete, bilateral or unilateral cleft lip and palate
  5. Intervention:Sonic toothbrush with activation of the dual light feature
  Interventions: Device: Toothbrush
- No surgery, Manual Toothbrush (Experimental): 1. Patient of record of the Craniofacial and Special Care Orthodontic Clinic at Children's Hospital Los Angeles
  2. Between the ages of 6 and 20 years
  3. Physical status of ASA I or II
  4. Diagnosis of craniofacial and/or isolated, complete or incomplete, bilateral or unilateral cleft lip and palate 5, Intervention:Manual toothbrush.
  Interventions: Device: Toothbrush
- No Surgery, Sonic Toothbrush (Experimental): 1. Patient of record of the Craniofacial and Special Care Orthodontic Clinic at Children's Hospital Los Angeles
  2. Between the ages of 6 and 20 years
  3. Physical status of ASA I or II
  4. Diagnosis of craniofacial and/or isolated, complete or incomplete, bilateral or unilateral cleft lip and palate
  5. Intervention:Sonic toothbrush without activation of the dual light feature.
  Interventions: Device: Toothbrush
- No Surgery, Sonic and Dual-light Toothbrush (Experimental): 1. Patient of record of the Craniofacial and Special Care Orthodontic Clinic at Children's Hospital Los Angeles
  2. Between the ages of 6 and 20 years
  3. Physical status of ASA I or II
  4. Diagnosis of craniofacial and/or isolated, complete or incomplete, bilateral or unilateral cleft lip and palate
  5. Intervention:Sonic toothbrush with activation of the dual light feature
  Interventions: Device: Toothbrush

INTERVENTIONS:
Device: Toothbrush — We will test three toothbrushes in patients undergoing surgery and a control no surgery group. These toothbrushes are manual toothbrushes, sonic toothbrushes, and sonic and dual light toothbrushes.

SUMMARY:
The study is a randomized clinical trial to compare the effectiveness of a dual light ultrasonic toothbrush on periodontal health in orthodontic patients undergoing surgery.

Patients with cleft lip and palate undergo bone graft and orthognathic surgery. The study will compare the periodontal outcomes in patients who use these toothbrushes during the post-surgical period.

DETAILED DESCRIPTION:
Pilot Study, Randomized Control Clinical Trial, study groups 1) Craniofacial and/or unilateral and bilateral cleft palate patients undergoing orthognathic surgery . 2) Craniofacial and/or unilateral and bilateral cleft palate patients undergoing bone-graft surgery 3) Craniofacial and/or unilateral and bilateral cleft palate patients with no pending surgery. Three Investigational device include Dual Light Therapy Sonic Toothbrush (BristlTM Toothbrush), Sonic Toothbrush(BRistlTM) and manual toothbrush to target disease gingivitis in 189 patients. Categorical variables scored from Plaque Index and Gingival Index will be analyzed using Fisher exact test and McNemar test. Parametric methods will be used to analyze data from Bleeding on Probing and Periodontal Probing Depth. To determine differences between groups and within each test at all time points, Student t-test will be used.

ELIGIBILITY:
Inclusion Criteria:

* Patient of record of the Craniofacial and Special Care Orthodontic Clinic at Children's Hospital Los Angeles
* Between the ages of 6 and 20 years
* Physical status of ASA I or II
* Diagnosis of craniofacial and/or isolated, complete or incomplete, bilateral or unilateral cleft lip and palate

Exclusion Criteria:

* physical inability to brush teeth
* cognitive inability to comprehend and follow directions.

Ages: 6 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 198 (Estimated)
Dates: Start 2024-03-11 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Löe and Silness Gingival Index | 18 weeks, 6 weeks apart evaluations
  This involves a two-step process: Step One (1): evaluation of the clinical appearance of the gingival tissue; and Step Two (2): assessment of inflammation based on induction of bleeding from probing11. Step One will not be accomplished chairside but will be measured using photographs; Step Two will be done chairside.
Bleeding index | 18 weeks, 6 weeks apart evaluations
  For Bleeding Index (Appendix IIC) and measurement of Probing Depth, the scorers will be calibrated following the Examiner Guide to Measuring Periodontal Parameters & Indices11. Probing Depth will be measured using a University of North Carolina (UNC) #15 manual probe and a #5 mouth mirror

SECONDARY OUTCOMES:
Turesky et al Modified Quigley-Hein Plaque Index and Modified Plaque Index for Orthodontic Patient | 18 weeks, 6 week apart evaluations
  After placement of five drops of Trace® plaque disclosing liquid under the tongue, the participant will swish the solution for 30 seconds. Upon expectoration, the participant will rinse his/her mouth with water three times. Immediately, intraoral photographs will be made. All photos for Gingival Index and Plaque Index will be scored by two blinded scorers with inter-rater reliability calculated. All scoring data will be assessed by statistician.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Yen, DMD, PhD, Principal Investigator — Children's Hospital Los Angeles and USC
Locations (1):
- Chilldren's Hospital Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ccahuana-Vasquez RA, Conde E, Grender JM, Cunningham P, Qaqish J, Goyal CR. An Eight-Week Clinical Evaluation of an Oscillating-Rotating Power Toothbrush with a Brush Head Utilizing Angled Bristles Compared with a Sonic Toothbrush in the Reduction of Gingivitis and Plaque. J Clin Dent. 2015;26(3):80-5. PMID 26665291